CLINICAL TRIAL: NCT03431376
Title: Potato Consumption Is Prospectively Associated With Risk of Hypertension: An 11.3-year Longitudinal Cohort Study
Brief Title: Potato Consumption and Risk of Hypertension
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Yu Zhang, Professor, Zhejiang University
Other Study IDs: Potato-CHNS-Cohort
Record Dates: First submitted 2018-02-02; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Hypertension
Keywords: potato consumption; hypertension; CHNS
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Government has popularized potatoes as a major staple food in China. Potato, a potassium-rich food with high glycemic responses after consumption, exhibits unclear effects on hypertension. In this study, the investigators aimed to examine the association between potato consumption and hypertension risk among Chinese people.

DETAILED DESCRIPTION:
Potato is considered as a superior crop due to its significant nutritive value and great production yield. China is the largest potato producer with a quarter of world production, followed by India, Russia, and USA. The potato production as well as consumption has enhanced in developing countries while continuously declined in developed countries during the last decade. The investigators therefore explored the prospective associations of consumption of total potatoes, sweet potatoes, stir-fried potatoes, and non stir-fried potatoes with the risk of hypertension in general people of the China Health and Nutrition Survey (CHNS) cohort study from 1989 to 2011. A total of 11,763 participants (≥20 years old) who were free of hypertension at baseline were enrolled from CHNS Cohort study. Cox proportional hazards regression models were used to estimate the associations after adjusting for potential confounders. This study provides new evidence on the association of various potato consumption with the incidence of hypertension in China. As urbanization accelerates across the whole domain of China, the tendency of transition to Western-style diets and lifestyles appears continuously and steeply growing. More and more potatoes will be consumed as processed potato products including potatoes chips and French fries, which may be a potential risk factor of hypertension occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-93 with complete data on diet and follow-up time
* Adults with no chronic disease history

Exclusion Criteria:

* Adults aged < 20 years
* Identified to be pregnant
* Previously diagnosed with hypertension, cancers, infarction, apoplexy, and diabetes

Ages: 20 Years to 93 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Of the 11,763 participants, 5,344 male and 6,419 female were enrolled, ranging from 20 to 93 years old. People who consumed the potatoes, sweet potatoes, stir-fried potatoes, and non stir-fried potatoes accounted for 57.3%, 15.0%, 51.8%, and 28.1%, respectively. There were about 90.4% people who consumed the potatoes through the stir-frying method.
Sampling Method: Probability Sample
Enrollment: 11763 (Actual)
Dates: Start 1989-01-01 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Hypertension | From entry into the study (baseline: 1989-2009) until 2011
  Incidence of hypertension, on basis of self-reported physician diagnosis, systolic blood pressure ≥ 140 mm Hg, diastolic blood pressure ≥ 90 mm Hg, or previous diagnose of hypertension by a physician or current use of anti-hypertensive drugs

SECONDARY OUTCOMES:
Potato consumption | From entry into the study (baseline: 1989-2009) until 2011
  The frequency and the quantity of daily average consumption of total potatoes, sweet potatoes, stir-fried potatoes, and non stir-fried potatoes (g/day) based on 3-day 24-hr recall

CONTACTS AND LOCATIONS:
Overall Officials: Jingjing Jiao, PhD, Study Director — Zhejiang University